CLINICAL TRIAL: NCT00609492
Title: Safety, Reactogenicity and Immunogenicity Following Booster Dose of GSK Biologicals´ Pneumococcal Conjugate Vaccine When Co-administered With a Booster Dose of Infanrix-IPV/Hib in Preterm Born Children at 16-18 Months of Age
Brief Title: Evaluate Safety and Immunogenicity of a Booster Dose of Pneumococcal Conjugate Vaccine in Preterm Born Infants.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109621; 2007-000596-42 (EudraCT Number)
Record Dates: First submitted 2008-01-25; First posted 2008-02-07 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Infections, Streptococcal; Streptococcus Pneumoniae Vaccines
MeSH Terms: conditions — Streptococcal Infections

ARMS (3):
- Preterm I Group (Experimental): Children born after a gestation period of 27-30 weeks
  Interventions: Biological: GSK Biologicals´ Pneumococcal Conjugate Vaccine (GSK1024850A); Biological: Infanrix™-IPV/Hib
- Preterm II Group (Experimental): Children born after a gestation period of 31-36 weeks
  Interventions: Biological: GSK Biologicals´ Pneumococcal Conjugate Vaccine (GSK1024850A); Biological: Infanrix™-IPV/Hib
- Full term Group (Active Comparator): Children born after a gestation period of more than 36 weeks
  Interventions: Biological: GSK Biologicals´ Pneumococcal Conjugate Vaccine (GSK1024850A); Biological: Infanrix™-IPV/Hib

INTERVENTIONS:
Biological: GSK Biologicals´ Pneumococcal Conjugate Vaccine (GSK1024850A) — Single dose, intramuscular injection
Biological: Infanrix™-IPV/Hib — Single dose, intramuscular injection

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity and immunogenicity of a booster dose of GlaxoSmithKline (GSK) Biologicals´ pneumococcal conjugate vaccine co-administered with a booster dose of DTPa-IPV/Hib (Infanrix-IPV/Hib) in preterm born children at the age of 16-18 months. This protocol posting deals with objectives & outcome measures of the booster phase. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT number =NCT00390910 ). Subjects participating in this study should have received three doses of pneumococcal vaccine in the primary study.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including, 16-18 months of age at the time of the booster vaccination.
* A male or female who previously participated in study 107737 and received three doses of pneumococcal conjugate vaccine.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Concurrently participating in another clinical study, at any time during the study period (active phase and extended safety follow-up), in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the booster dose of study vaccines, or planned use during the study period (active phase and 5 months extended safety follow-up).
* Chronic administration of immunosuppressants or other immune-modifying drugs within 6 months prior to the booster dose of study vaccine.
* Planned administration/administration of a vaccine not foreseen by the study protocol, during the period starting from one month (30 days) before the booster dose of study vaccines (Visit 1) and up to the follow-up visit (Visit 2).
* Previous vaccination against diphtheria, tetanus, pertussis, polio, hepatitis B, Haemophilus influenzae type b and/or Streptococcus pneumoniae other than the study vaccines from study 107737
* History of or intercurrent diphtheria, tetanus, hepatitis B, pertussis, polio, Haemophilus influenzae type b disease.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* History of seizures or progressive neurological disease
* Acute disease at the time of enrolment.
* Febrile illness defined as oral, axillary or tympanic temperature < 37.5°C / rectal temperature < 38°C. A temperature greater than or equal to these cut-offs warrants deferral of the vaccination pending recovery of the subject.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* Administration of immunoglobulins, with the exception of monoclonal antibodies against RSV, and/or any blood products within three months preceding the booster dose of study vaccines or planned administration during the active phase of the study.

Ages: 16 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 245 (Actual)
Dates: Start 2008-01-03 (Actual); Primary Completion 2008-11-10 (Actual); Study Completion 2009-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Ioannina
  - GSK Investigational Site, Thessaloniki
- Spain (3):
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Móstoles/Madrid

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=255

REFERENCES:
- [Background] Omenaca F, Merino JM, Tejedor JC, Constantopoulos A, Papaevangelou V, Kafetzis D, Tsirka A, Athanassiadou F, Anagnostakou M, Francois N, Borys D, Schuerman L. Immunization of preterm infants with 10-valent pneumococcal conjugate vaccine. Pediatrics. 2011 Aug;128(2):e290-8. doi: 10.1542/peds.2010-1184. Epub 2011 Jul 4. PMID 21727108
- [Background] Omenaca F et al. Booster vaccination of preterm-born children with 10-valent pneumococcal non-typeable haemophilus influenzae protein D-conjugate vaccine (PHiD-CV): antibody responses and safety. Abstract presented at the 6th World Congress of the World Society for Pediatric Infectious Diseases (WSPID). Beunos Aires, Argentina, 18-22 November 2009.
- [Background] Omenaca F et al. Immunogenicity and safety of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) following primary and booster vaccination in preterm-born children. Abstract presented at Excellence In Paediatrics. Florence, Italy, 3-6 December 2009.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 109621 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109621 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109621 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109621 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109621 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109621 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109621 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Preterm I Group: Children born after a gestation period of 27-30 weeks (189-216 days) who were previously vaccinated with three primary doses of Synflorix™ vaccine co-administered with Infanrix Hexa™ in study 10PN-PD-DIT-015 (107737), additionally received one booster dose of Synflorix™ vaccine co-administered with a single dose of Infanrix™-IPV/Hib vaccine, intramuscularly in the deltoid/thigh, at 16-18 months of age.
- Preterm II Group: Children born after a gestation period of 31-36 weeks (217-258 days) who were previously vaccinated with three primary doses of Synflorix™ vaccine co-administered with Infanrix Hexa™ in study 10PN-PD-DIT-015 (107737), additionally received one booster dose of Synflorix™ vaccine co-administered with a single dose of Infanrix™-IPV/Hib vaccine, intramuscularly in the deltoid/thigh, at 16-18 months of age.
- Full Term Group: Children born after a gestation period of more than 36 weeks (more than 258 days) who were previously vaccinated with three primary doses of Synflorix™ vaccine co-administered with Infanrix Hexa™ in study 10PN-PD-DIT-015 (107737), additionally received one booster dose of Synflorix™ vaccine co-administered with a single dose of Infanrix™-IPV/Hib vaccine, intramuscularly in the deltoid/thigh, at 16-18 months of age.
Period: Overall Study
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Started | 44 | 72 | 129
Completed | 43 | 69 | 122
Not Completed | 1 | 3 | 7
Not completed — Withdrawal by Subject | 0 | 2 | 3
Not completed — Lost to Follow-up | 1 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group | Total
Number analyzed (Participants) | 44 | 72 | 129 | 245
Age, Continuous [Mean (Standard Deviation); unit: Months] | 16.8 (0.63) | 17.2 (0.68) | 16.6 (0.73) | 16.81 (0.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 29 | 50 | 95
  Male | 28 | 43 | 79 | 150

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Fever With Rectal Temperature Above (>) 39.0 Degrees Celsius (°C)
Description: Fever was measured as rectal temperature. Assessment of occurrences of fever > 39.0 °C was performed within 4-days (Day 0-3) after booster vaccination of Synflorix™ and Infanrix™-IPV/Hib vaccine.
Time Frame: Within 4-days (Day 0-3) after booster vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available and who had filled in the symptom sheet.
Measure: Number; unit: Subjects
Groups:
- Preterm Group: Pooled group with subjects from the Preterm I Group and the Preterm II Group who were previously vaccinated with three primary doses of Synflorix™ vaccine co-administered with Infanrix Hexa™ in study 10PN-PD-DIT-015 (107737), additionally received one booster dose of Synflorix™ vaccine co-administered with a single dose of Infanrix™-IPV/Hib vaccine, intramuscularly in the deltoid/thigh, at 16-18 months of age.
Arm/Group | Preterm Group | Full Term Group
Number analyzed (Participants) | 112 | 122
Subjects | 8 | 6

2. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed included pain, redness and swelling. Grade 3 pain was defined as crying when limb was moved/spontaneously painful. Grade 3 swelling/redness was defined as swelling/redness larger than (>) 30 millimeters (mm). "Any" is defined as incidence of the specified symptom regardless of intensity.
Time Frame: Within 4-days (Day 0-3) after booster vaccination
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Preterm Group | Full Term Group
Number analyzed (Participants) | 112 | 122
Subjects
  Any Pain | 47 | 67
  Grade 3 Pain | 5 | 4
  Any Redness | 35 | 65
  Grade 3 Redness | 3 | 19
  Any Swelling | 27 | 55
  Grade 3 Swelling | 1 | 14

3. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited General Symptoms
Description: Solicited general symptoms assessed included drowsiness, fever (defined as rectal temperature ≥ 38.0°C), irritability, and loss of appetite. Grade 3 drowsiness was defined as drowsiness which prevented normal everyday activities. Grade 3 fever was defined as fever (rectal temperature) above (>) 40.0 degree Celsius (°C). Grade 3 irritability was defined as crying that could not be comforted/preventing normal activity. Grade 3 loss of appetite was defined as the subject not eating at all. "Any" is defined as incidence of the specified symptom regardless of intensity or relationship to study vaccination.
Time Frame: Within 4-days (Day 0-3) after booster vaccination
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Preterm Group | Full Term Group
Number analyzed (Participants) | 112 | 122
Subjects
  Any Drowsiness | 21 | 33
  Grade 3 Drowsiness | 1 | 1
  Any Fever | 34 | 39
  Grade 3 Fever | 0 | 1
  Any Irritability | 36 | 49
  Grade 3 Irritability | 2 | 2
  Any Loss of appetite | 26 | 35
  Grade 3 Loss of appetite | 0 | 1

4. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. "Any" is defined as incidence of an unsolicited AE regardless of intensity or relationship to study vaccination.
Time Frame: Within 31-days (Day 0-30) after booster vaccination
Population: The analysis was performed on the Total vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Preterm Group | Full Term Group
Number analyzed (Participants) | 116 | 129
Subjects | 17 | 24

5. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Throughout the active phase of the study (Month 0 to Month 1)
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Preterm Group | Full Term Group
Number analyzed (Participants) | 116 | 129
Subjects | 0 | 0

6. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 5
Time Frame: Throughout the entire study period starting from Month 0 up to the end of the extended safety follow-up (Month 6)
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Preterm Group | Full Term Group
Number analyzed (Participants) | 116 | 129
Subjects | 3 | 1

7. Secondary Outcome: Number of Seropositive Subjects for Anti-pneumococcal Serotypes
Description: A seropositive subject was defined as a subject who had the anti-pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C , 19F and 23F concentrations greater than or equal to (≥) the cut-off value of 0.05 micrograms per milliliter (μg/mL).
Time Frame: Prior to (Pre-booster) and one month after (Post-booster) the administration of the booster dose of Synflorix™ vaccine co-administered with the booster dose of Infanrix™ -IPV/Hib vaccine
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Number; unit: Subjects
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 43 | 69 | 125
Subjects
  Anti-1, Pre-booster [N=43;66;121] | 39 | 56 | 111
  Anti-1, Post-booster [N=43;66;119] | 43 | 66 | 119
  Anti-4, Pre-booster [N=43;69;123] | 40 | 68 | 120
  Anti-4, Post-booster [N=43;66;119] | 43 | 66 | 119
  Anti-5, Pre-booster [N=43;68;124] | 41 | 66 | 122
  Anti-5, Post-booster [N=43;66;119] | 43 | 66 | 119
  Anti-6B, Pre-booster [N=43;67;124] | 41 | 66 | 119
  Anti-6B, Post-booster [N=42;66;119] | 42 | 65 | 119
  Anti-7F, Pre-booster [N=43;65;123] | 42 | 65 | 123
  Anti-7F, Post-booster [N=43;66;118] | 43 | 66 | 118
  Anti-9V, Pre-booster [N=43;69;123] | 43 | 69 | 123
  Anti-9V, Post-booster [N=43;66;119] | 43 | 66 | 119
  Anti-14, Pre-booster [N=43;68;124] | 43 | 68 | 121
  Anti-14, Post-booster [N=43;66;119] | 43 | 66 | 119
  Anti-18C, Pre-booster [N=43;68;125] | 43 | 68 | 123
  Anti-18C, Post-booster [N=43;66;119] | 43 | 66 | 118
  Anti-19F, Pre-booster [N=43;68;125] | 43 | 68 | 125
  Anti-19F, Post-booster [N=43;66;119] | 43 | 66 | 119
  Anti-23F, Pre-booster [N=43;69;123] | 41 | 68 | 122
  Anti-23F, Post-booster [N=42;66;119] | 41 | 66 | 118

8. Secondary Outcome: Number of Seroprotected Subjects Against Anti-pneumococcal Serotypes
Description: A seroprotected subjects was defined as a subject who had anti-pneumococcal serotypes antibody concentrations greater than or equal to (≥) the threshold value of 0.20 micrograms per milliliter (μg/mL). The anti-pneumococcal serotypes assessed were 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F.
Time Frame: Prior to (Pre-booster) and one month after (Post-booster) the administration of the booster dose of Synflorix™ vaccine co-administered with the booster dose of Infanrix™-IPV/Hib vaccine
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Number; unit: Subjects
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 44 | 69 | 125
Subjects
  Anti-1, Pre-booster [N=43;66;121] | 16 | 28 | 53
  Anti-1, Post-booster [N=43;66;119] | 43 | 66 | 118
  Anti-4, Pre-booster [N=43;69;123] | 23 | 40 | 82
  Anti-4, Post-booster [N=43;66;119] | 43 | 66 | 119
  Anti-5, Pre-booster [N=43;68;124] | 27 | 43 | 105
  Anti-5, Post-booster [N=43;66;119] | 43 | 66 | 119
  Anti-6B, Pre-booster [N=43;67;124] | 28 | 41 | 99
  Anti-6B, Post-booster [N=42;66;119] | 42 | 65 | 119
  Anti-7F, Pre-booster [N=43;65;123] | 34 | 56 | 115
  Anti-7F, Post-booster [N=43;66;118] | 43 | 66 | 118
  Anti-9V, Pre-booster [N=43;69;123] | 39 | 59 | 115
  Anti-9V, Post-booster [N=43;66;119] | 43 | 66 | 119
  Anti-14, Pre-booster [N=43;68;124] | 41 | 55 | 105
  Anti-14, Post-booster [N=43;66;119] | 43 | 66 | 119
  Anti-18C, Pre-booster [N=43;68;125] | 36 | 60 | 106
  Anti-18C, Post-booster [N=43;66;119] | 43 | 66 | 118
  Anti-19F, Pre-booster [N=43;68;125] | 38 | 66 | 120
  Anti-19F, Post-booster [N=43;66;119] | 43 | 66 | 119
  Anti-23F, Pre-booster [N=43;69;123] | 30 | 45 | 99
  Anti-23F, Post-booster [N=42;66;119] | 41 | 66 | 118

9. Secondary Outcome: Antibody Concentrations Against Pneumococcal Serotypes
Description: Seropositivity status was defined as the anti-pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody concentrations greater than or equal to (≥) the cut-off value of 0.05 micrograms per milliliter (µg/mL). Antibody concentrations were measured by 22F enzyme-linked immunosorbent assay (ELISA), presented as geometric mean concentrations (GMCs).
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 43 | 69 | 125
µg/mL
  Anti-1, Pre-booster [N=43;66;121] | 0.15 [0.11 to 0.2] | 0.14 [0.11 to 0.18] | 0.17 [0.15 to 0.21]
  Anti-1, Post-booster [N=43;66;119] | 1.57 [1.20 to 2.05] | 1.74 [1.41 to 2.15] | 1.98 [1.66 to 2.37]
  Anti-4, Pre-booster [N=43;69;123] | 0.25 [0.18 to 0.35] | 0.24 [0.20 to 0.30] | 0.30 [0.25 to 0.35]
  Anti-4, Post-booster [N=43;66;119] | 2.98 [2.31 to 3.85] | 3.67 [3.07 to 4.39] | 4.23 [3.67 to 4.88]
  Anti-5, Pre-booster [N=43;68;124] | 0.24 [0.18 to 0.33] | 0.27 [0.21 to 0.34] | 0.40 [0.34 to 0.48]
  Anti-5, Post-booster [N=43;66;119] | 1.84 [1.43 to 2.38] | 2.38 [1.93 to 2.94] | 2.58 [2.20 to 3.02]
  Anti-6B, Pre-booster [N=43;67;124] | 0.28 [0.21 to 0.38] | 0.30 [0.23 to 0.37] | 0.37 [0.31 to 0.45]
  Anti-6B, Post-booster [N=42;66;119] | 2.44 [1.87 to 3.17] | 2.46 [1.97 to 3.06] | 2.67 [2.27 to 3.13]
  Anti-7F, Pre-booster [N=43;65;123] | 0.42 [0.31 to 0.56] | 0.46 [0.37 to 0.58] | 0.66 [0.57 to 0.77]
  Anti-7F, Post-booster [N=43;66;118] | 3.11 [2.48 to 3.90] | 4.16 [3.52 to 4.90] | 3.93 [3.45 to 4.47]
  Anti-9V, Pre-booster [N=43;69;123] | 0.51 [0.39 to 0.67] | 0.42 [0.35 to 0.52] | 0.59 [0.51 to 0.69]
  Anti-9V, Post-booster [N=43;66;119] | 2.87 [2.23 to 3.70] | 3.47 [2.86 to 4.20] | 4.17 [3.60 to 4.83]
  Anti-14, Pre-booster [N=43;68;124] | 0.78 [0.54 to 1.11] | 0.48 [0.37 to 0.61] | 0.68 [0.55 to 0.84]
  Anti-14, Post-booster [N=43;66;119] | 4.88 [3.42 to 6.98] | 5.14 [4.22 to 6.25] | 5.98 [5.10 to 7.02]
  Anti-18C, Pre-booster [N=43;68;125] | 0.58 [0.42 to 0.80] | 0.56 [0.45 to 0.70] | 0.60 [0.49 to 0.73]
  Anti-18C, Post-booster [N=43;66;119] | 9.51 [7.36 to 12.29] | 13.20 [10.97 to 15.89] | 12.38 [10.21 to 15.00]
  Anti-19F, Pre-booster [N=43;68;125] | 0.86 [0.58 to 1.30] | 1.07 [0.78 to 1.46] | 1.27 [1.02 to 1.59]
  Anti-19F, Post-booster [N=43;66;119] | 6.83 [5.24 to 8.89] | 9.78 [8.19 to 11.68] | 9.72 [8.38 to 11.29]
  Anti-23F, Pre-booster [N=43;69;123] | 0.27 [0.20 to 0.36] | 0.30 [0.24 to 0.38] | 0.42 [0.35 to 0.51]
  Anti-23F, Post-booster [N=42;66;119] | 2.70 [1.91 to 3.81] | 3.45 [2.93 to 4.06] | 3.30 [2.74 to 3.99]

10. Secondary Outcome: Number of Seropositive Subjects for Pneumococcal Cross-reactive Serotypes 6A and 19A
Description: A seropositive subject was defined as a subject who had the anti-pneumococcal serotypes 6A and 19A concentrations greater than or equal to (≥) the cut-off value of 0.05 micrograms per milliliter (μg/mL).
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 43 | 67 | 122
Subjects
  Anti-6A, Pre-booster [N=42;67;122] | 34 | 51 | 98
  Anti-6A, Post-booster [N=42;66;118] | 41 | 63 | 115
  Anti-19A, Pre-booster [N=43;67;121] | 28 | 49 | 95
  Anti-19A, Post-booster [N=42;66;118] | 40 | 63 | 113

11. Secondary Outcome: Antibody Concentrations Against Pneumococcal Cross-reactive Serotypes 6A and 19A
Description: Seropositivity status was defined as the anti-pneumococcal cross-reactive serotypes 6A and 19A antibody concentrations greater than or equal to (≥) the cut-off value of 0.05 micrograms per milliliter (µg/mL). Antibody concentrations were measured by 22F enzyme-linked immunosorbent assay (ELISA), presented as geometric mean concentrations (GMCs).
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 43 | 67 | 122
µg/mL
  Anti-6A, Pre-booster [N=42;67;122] | 0.12 [0.08 to 0.17] | 0.12 [0.09 to 0.16] | 0.14 [0.12 to 0.18]
  Anti-6A, Post-booster [N=42;66;118] | 0.70 [0.47 to 1.05] | 0.77 [0.55 to 1.07] | 0.79 [0.61 to 1.02]
  Anti-19A, Pre-booster [N=43;67;121] | 0.14 [0.08 to 0.24] | 0.15 [0.10 to 0.22] | 0.16 [0.12 to 0.22]
  Anti-19A, Post-booster [N=42;66;118] | 0.65 [0.40 to 1.04] | 0.93 [0.64 to 1.37] | 1.10 [0.82 to 1.47]

12. Secondary Outcome: Number of Seropositive Subjects for Protein D Antibodies (Anti-PD)
Description: A seropositive subject was defined as a subject who had anti-PD concentration greater than or equal to (≥) the value of 100 ELISA units per milliliter (EL.U/mL).
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 43 | 67 | 123
Subjects
  Anti-PD, Pre-booster [N=42;67;123] | 39 | 58 | 114
  Anti-PD, Post-booster [N=43;66;118] | 43 | 66 | 117

13. Secondary Outcome: Antibody Concentrations Against Protein D (Anti-PD)
Description: Seropositivity status was defined as the anti-protein D (Anti-PD) antibody concentrations greater than or equal to (≥) 100 ELISA units per milliliter (EL.U/mL). Antibody concentrations were measured by enzyme-linked immunosorbent assay (ELISA), presented as geometric mean concentrations (GMCs).
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 43 | 67 | 123
EL.U/mL
  Anti-PD, Pre-booster [N=42;67;123] | 478.3 [361.4 to 633.1] | 340.0 [258.1 to 447.9] | 383.7 [317.6 to 463.5]
  Anti-PD, Post-booster [N=43;66;118] | 1892.9 [1415.1 to 2532.2] | 1576.5 [1232.7 to 2016.1] | 1533.6 [1278.2 to 1840.1]

14. Secondary Outcome: Number of Seroprotected Subjects Against Anti-diphtheria (Anti-DT) and Anti-tetanus Toxoids (Anti-TT)
Description: A seroprotected subject was defined as a subject who had anti-DT and anti-TT concentrations greater than or equal to (≥) the value of 0.1 international units per milliliter (IU/mL).
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 23 | 34 | 60
Subjects
  Anti-DT, Pre-booster [N=23;31;59] | 20 | 27 | 51
  Anti-DT, Post-booster [N=21;34;60] | 21 | 34 | 60
  Anti-TT, Pre-booster [N=23;32;59] | 23 | 32 | 59
  Anti-TT, Post-booster [N=21;34;60] | 21 | 34 | 60

15. Secondary Outcome: Antibody Concentrations Against Anti-diphtheria (Anti-DT) and Anti-tetanus Toxoids (Anti-TT)
Description: Seropositivity status was defined as the anti-diphtheria toxoid (Anti-DT) and anti-tetanus toxoid (Anti-TT) antibody concentrations greater than or equal to (≥) 0.1 international units per milliliter (IU/mL). Antibody concentrations were measured by enzyme-linked immunosorbent assay (ELISA), presented as geometric mean concentrations (GMCs).
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 23 | 34 | 60
IU/mL
  Anti-DT, Pre-booster [N=23;31;59] | 0.381 [0.210 to 0.689] | 0.674 [0.380 to 1.196] | 0.481 [0.324 to 0.716]
  Anti-DT, Post-booster [N=21;34;60] | 6.252 [4.572 to 8.551] | 9.982 [7.392 to 13.478] | 6.730 [5.254 to 8.620]
  Anti-TT, Pre-booster [N=23;32;59] | 0.821 [0.591 to 1.141] | 0.726 [0.601 to 0.877] | 0.918 [0.711 to 1.184]
  Anti-TT, Post-booster [N=21;34;60] | 12.374 [9.629 to 15.903] | 14.392 [11.717 to 17.676] | 13.026 [11.176 to 15.183]

16. Secondary Outcome: Number of Seroprotected Subjects Against Anti-polyribosyl-ribitol Phosphate (Anti-PRP)
Description: A seroprotected subject was defined as a subject who had anti-PRP concentrations greater than or equal to (≥) the value of 0.15 micrograms per milliliter (µg /mL).
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 23 | 34 | 59
Subjects
  Anti-PRP, Pre-booster [N=23;32;59] | 16 | 26 | 50
  Anti-PRP, Post-booster [N=20;34;59] | 20 | 34 | 59

17. Secondary Outcome: Number of Subjects With Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibody Concentration ≥ 1.0 µg/mL
Description: The concentration of anti-polyribosyl-ribitol phosphate (Anti-PRP) antibody assessed was greater than or equal to (≥) the value of 1.0 micrograms per milliliter (µg /mL).
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 23 | 34 | 59
Subjects
  Anti-PRP, Pre-booster [N=23;32;59] | 6 | 9 | 20
  Anti-PRP, Post-booster [N=20;34;59] | 20 | 34 | 59

18. Secondary Outcome: Antibody Concentrations Against Anti-polyribosyl-ribitol-phosphate (Anti-PRP)
Description: Seropositivity status was defined as the anti-polyribosyl-ribitol-phosphate (Anti-PRP) antibody concentrations greater than or equal to (≥) 0.15 micrograms per milliliter (µg /mL) and ≥ 1.0 µg/mL. Antibody concentrations were measured by enzyme-linked immunosorbent assay (ELISA), presented as geometric mean concentrations (GMCs).
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 23 | 34 | 59
µg/mL
  Anti-PRP, Pre-booster [N=23;32;59] | 0.376 [0.196 to 0.719] | 0.509 [0.312 to 0.832] | 0.577 [0.372 to 0.896]
  Anti-PRP, Post-booster [N=20;34;59] | 33.731 [17.907 to 63.540] | 36.902 [25.148 to 54.148] | 38.713 [27.736 to 54.034]

19. Secondary Outcome: Number of Seropositive Subjects for Anti-pertussis Toxoid (Anti-PT), Anti- Filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN)
Description: A seropositive subject was defined as a subject who had anti-PT, anti-FHA and anti-PRN concentrations greater than or equal to (≥) the value of 5 ELISA units per milliliter (EL.U/mL).
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 23 | 34 | 60
Subjects
  Anti-PT, Pre-booster [N=22;32;58] | 10 | 11 | 30
  Anti-PT, Post-booster [N=21;34;59] | 21 | 34 | 59
  Anti-FHA, Pre-booster [N=20;27;47] | 19 | 24 | 43
  Anti-FHA, Post-booster [N=21;34;59] | 21 | 34 | 59
  Anti-PRN, Pre-booster [N=23;32;59] | 20 | 28 | 47
  Anti-PRN, Post-booster [N=21;34;60] | 21 | 34 | 60

20. Secondary Outcome: Antibody Concentrations Against Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN)
Description: Seropositivity status was defined as the anti-pertussis toxoid (Anti-PT), anti-filamentous haemagglutinin (Anti-FHA) and anti-pertactin (Anti-PRN) antibody concentrations greater than or equal to (≥) 5 ELISA units per milliliter (EL.U /mL). Antibody concentrations were measured by enzyme-linked immunosorbent assay (ELISA), presented as geometric mean concentrations (GMCs).
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 23 | 34 | 60
EL.U/mL
  Anti-PT, Pre-booster [N=22;32;58] | 5.7 [3.3 to 9.8] | 3.8 [3.0 to 4.7] | 5.5 [4.4 to 6.9]
  Anti-PT, Post-booster [N=21;34;59] | 38.4 [29.8 to 49.5] | 32.7 [24.2 to 44.2] | 45.1 [37.0 to 54.9]
  Anti-FHA, Pre-booster [N=20;27;47] | 39.4 [18.4 to 84.2] | 13.7 [9.3 to 20.1] | 17.0 [12.4 to 23.3]
  Anti-FHA, Post-booster [N=21;34;59] | 250.3 [162.4 to 385.8] | 275.3 [207.0 to 366.1] | 229.0 [188.1 to 278.9]
  Anti-PRN, Pre-booster [N=23;32;59] | 16.7 [9.4 to 29.9] | 10.3 [7.4 to 14.2] | 11.3 [8.7 to 14.8]
  Anti-PRN, Post-booster [N=21;34;60] | 259.7 [151.5 to 445.2] | 286.5 [192.6 to 426.0] | 264.5 [200.2 to 349.5]

21. Secondary Outcome: Number of Subjects With Vaccine Response for Anti-PT, Anti-FHA and Anti-PRN Antibodies
Description: Vaccine response was defined as antibody concentrations ≥ 5 EL.U/mL at post-booster, for initially seronegative subjects (S-) (with concentrations < 5 EL.U/mL) and for initially seropositive subjects (S+) (with concentrations ≥ 5 EL.U/mL), antibody concentrations at post-booster ≥ 2 fold the pre-vaccination antibody concentration.
Time Frame: One month after (Post-booster) the administration of the booster dose of Synflorix™ vaccine co-administered with the booster dose of Infanrix™-IPV/Hib vaccine
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 19 | 28 | 45
Subjects
  Anti-PT, S- [N=11;21;27] | 11 | 21 | 27
  Anti-PT, S+ [N=9;11;27] | 9 | 11 | 24
  Anti-FHA, S- [N=1;3;4] | 1 | 3 | 4
  Anti-FHA, S+ [N=17;24;39] | 17 | 24 | 37
  Anti-PRN, S- [N=2;4;11] | 2 | 4 | 11
  Anti-PRN, S+ [N=19;28;45] | 19 | 28 | 44

22. Secondary Outcome: Number of Seroprotected Subjects Against Anti-polio Type 1, 2 and 3 (Anti-Polio 1, 2 and 3)
Description: A seroprotected subject was defined as a subject who had anti-polio types 1, 2 and 3 titers greater than or equal to (≥) the value of 8.
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 17 | 29 | 53
Subjects
  Anti-Polio 1, Pre-booster [N=17;29;53] | 17 | 22 | 49
  Anti-Polio 1, Post-booster [N=3;8;20] | 3 | 8 | 20
  Anti-Polio 2, Pre-booster [N=17;29;53] | 17 | 26 | 47
  Anti-Polio 2, Post-booster [N=3;8;20] | 3 | 8 | 20
  Anti-Polio 3, Pre-booster [N=17;29;53] | 12 | 23 | 51
  Anti-Polio 3, Post-booster [N=3;8;20] | 3 | 8 | 20

23. Secondary Outcome: Antibody Titers Against Anti-polio Type 1, 2 and 3
Description: Seroprotection status was defined as the anti-polio type 1, anti-polio type 2 and anti-polio type 3 antibody titers greater than or equal to (≥) the cut-off value of 8, presented as geometric mean titers (GMTs).
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 17 | 29 | 53
Titers
  Anti-Polio 1, Pre-booster [N=17;29;53] | 52.3 [31.2 to 87.6] | 34.8 [19.4 to 62.7] | 54.7 [37.7 to 79.3]
  Anti-Polio 1, Post-booster [N=3;8;20] | 512.0 [115.3 to 2274.0] | 1386.7 [456.6 to 4210.9] | 1327.9 [795.4 to 2217.1]
  Anti-Polio 2, Pre-booster [N=17;29;53] | 65.2 [37.4 to 113.7] | 47.3 [26.2 to 85.3] | 50.9 [33.7 to 76.7]
  Anti-Polio 2, Post-booster [N=3;8;20] | 1290.1 [147.8 to 11259.3] | 2048.0 [759.7 to 5520.9] | 1116.9 [600.9 to 2076.1]
  Anti-Polio 3, Pre-booster [N=17;29;53] | 23.0 [10.0 to 53.2] | 31.3 [16.8 to 58.4] | 84.3 [59.0 to 120.4]
  Anti-Polio 3, Post-booster [N=3;8;20] | 574.7 [36.1 to 9148.9] | 1448.1 [464.0 to 4519.2] | 1692.5 [1147.7 to 2495.9]

24. Secondary Outcome: Antibody Concentrations Against Anti-hepatitis B Surface Antigen (HBs)
Description: Seroprotection status was defined as the Anti-HBs antibody concentrations greater than or equal to (≥) 10 milli international units per milliliter (mIU/mL), presented as geometric mean concentrations (GMCs).
Time Frame: Prior to (Pre-booster) the administration of the booster dose of Synflorix™ vaccine co-administered with the booster dose of Infanrix™-IPV/Hib vaccine
Population: The analysis was performed on the ATP cohort for persistence, which included all subjects for whom assay results were available for antibodies against at least one study vaccine antigen component for the blood sampling taken before the administration of the study booster dose.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 2 | 1 | 12
mIU/mL | 21.9 [1.9 to 246.8] | 117.2 [117.2 to 117.2] | 37.2 [15.6 to 88.8]

25. Secondary Outcome: Number of Seropositive Subjects for Opsonophagocytic Activity (OPA) Against Pneumococcal Serotypes
Description: A seropositive subject was defines as a subject with opsonophagocytic activity cut-off value greater than or equal to (≥) the value of 8. The vaccine pneumococcal serotypes investigated were 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F.
Time Frame: as for outcome 21
Population: as for outcome 7
Measure: Number; unit: Subjects
Groups:
- Preterm II Group: Children born after a gestation period of 31-36 weeks (217-258 days) who were previously vaccinated with three primary doses of Synflorix™ vaccine co-administered with Infanrix Hexa™ in study 10PN-PD-DIT-015 (107737), additionally received one booster dose of Synflorix™ vaccine co-administered with a single dose of Infanrix™-IPV/Hib vaccine, intramuscularly in the deltoid
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 38 | 55 | 100
Subjects
  OPA Anti-1, [N=37;52;99] | 34 | 49 | 93
  OPA Anti-4, [N=36;55;100] | 35 | 55 | 100
  OPA Anti-5, [N=34;50;93] | 32 | 48 | 92
  OPA Anti-6B, [N=35;51;98] | 33 | 49 | 92
  OPA Anti-7F, [N=37;49;99] | 37 | 49 | 99
  OPA Anti-9V, [N=38;47;100] | 38 | 47 | 100
  OPA Anti-14, [N=36;52;99] | 36 | 52 | 99
  OPA Anti-18C, [N=37;50;100] | 37 | 50 | 100
  OPA Anti-19F, [N=36;52;96] | 36 | 51 | 96
  OPA Anti-23F, [N=37;54;99] | 37 | 54 | 99

26. Secondary Outcome: Opsonophagocytic Activity (OPA) Against Pneumococcal Serotypes
Description: Seropositivity status was defined as the opsonophagocytic activity (OPA) against pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F, with a cut-off value greater than or equal to (≥) 8, presented as geometric mean titers (GMTs).
Time Frame: as for outcome 21
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 38 | 55 | 100
Titers
  OPA Anti-1, [N=37;52;99] | 125 [74.1 to 210.8] | 143.6 [93.1 to 221.3] | 170.9 [124.6 to 234.3]
  OPA Anti-4, [N=36;55;100] | 971.8 [623.7 to 1514.1] | 1307.2 [1070.0 to 1596.9] | 1479.3 [1259.6 to 1737.3]
  OPA Anti-5, [N=34;50;93] | 69.2 [45.0 to 106.4] | 120.0 [81.2 to 177.1] | 176.9 [138.1 to 226.5]
  OPA Anti-6B, [N=35;51;98] | 659.0 [353.9 to 1227.3] | 459.1 [286.7 to 735.3] | 635.0 [437.3 to 922.1]
  OPA Anti-7F, [N=37;49;99] | 6008.9 [4318.7 to 8360.5] | 4851.1 [3954.4 to 5951.1] | 4372.6 [3658.8 to 5225.5]
  OPA Anti-9V, [N=38;47;100] | 1666.4 [1218.1 to 2279.6] | 2192.5 [1724.3 to 2787.8] | 1798.8 [1522.8 to 2124.7]
  OPA Anti-14, [N=36;52;99] | 1489.5 [980.7 to 2262.3] | 1895.3 [1477.3 to 2431.7] | 1342.7 [1095.4 to 1646.0]
  OPA Anti-18C, [N=37;50;100] | 1656.0 [1005.6 to 2727.0] | 1672.4 [1154.4 to 2422.9] | 1561.9 [1251.2 to 1949.8]
  OPA Anti-19F, [N=36;52;96] | 379.3 [241.3 to 596.2] | 486.3 [327.9 to 721.3] | 626.8 [473.1 to 830.3]
  OPA Anti-23F, [N=37;54;99] | 2881.8 [1956.7 to 4244.3] | 2510.2 [2076.2 to 3035.0] | 3208.6 [2667.3 to 3859.8]

27. Secondary Outcome: Number of Seropositive Subjects for Opsonophagocytic Activity (OPA) Against Pneumococcal Cross-reactive Serotypes 6A and 19A
Description: A seropositive subject was defined as a subject with opsonophagocytic activity against pneumococcal cross-reactive serotypes 6A and 19A greater than or equal to (≥) the cut-off value of 8.
Time Frame: as for outcome 21
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 38 | 52 | 95
Subjects
  OPA Anti-6A, [N=34;50;95] | 31 | 45 | 79
  OPA Anti-19A, [N=38;52;95] | 23 | 30 | 56

28. Secondary Outcome: Opsonophagocytic Activity (OPA) Against Pneumococcal Cross-reactive Serotypes 6A and 19A
Description: Seropositivity status was defined as the opsonophagocytic activity (OPA) against pneumococcal cross-reactive serotypes 6A and 19A, with a cut-off value greater than or equal to (≥) 8, presented as geometric mean titers (GMTs).
Time Frame: as for outcome 21
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Preterm I Group | Preterm II Group | Full Term Group
Number analyzed (Participants) | 38 | 52 | 95
Titers
  OPA Anti-6A, [N=34;50;95] | 270.6 [152.9 to 478.6] | 218.2 [137.4 to 346.6] | 207.4 [136.8 to 314.4]
  OPA Anti-19A, [N=38;52;95] | 31.9 [16.0 to 63.6] | 41.4 [22.0 to 77.8] | 51.7 [32.1 to 83.5]

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-days (Day 0-3) post-booster vaccination. Unsolicited AEs: within 31-days (Day 0-30) post-booster vaccination; SAEs: throughout the entire study period starting from Month 0 up to the end of study.
Arm/Group | Preterm Group | Full Term Group
Serious Adverse Events (participants affected / at risk) | 3/116 | 1/129
Other Adverse Events (participants affected / at risk) | 71/116 | 98/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preterm Group (N=116) | Full Term Group (N=129)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0
Latent tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Preterm Group (N=116) | Full Term Group (N=129)
Pain (General disorders) | 47/112 (47) | 67/122 (67)
Redness (General disorders) | 35/112 (35) | 65/122 (65)
Swelling (General disorders) | 27/112 (27) | 55/122 (55)
Drowsiness (General disorders) | 21/112 (21) | 33/122 (33)
Fever (rectal temperature measurement) (General disorders) | 34/112 (34) | 39/122 (39)
Irritability (General disorders) | 36/112 (36) | 49/122 (49)
Loss of appetite (General disorders) | 26/112 (26) | 35/122 (35)

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.